CLINICAL TRIAL: NCT06224465
Title: Effect of Anti-aging Therapy on Fitness Enhancement in Perimenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Suzy Samih Nazmy, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005035
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Aging Well
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: intervention: aerobic exercises: walking :30 min on treadmill 30min at least three times per week for 12 weeks 2)Muscle strength Exercises: For upper extremity : hand grip exercise, arm flexion exercise ten repetition for each exercise three times per week.
  Theraband exercises for upper limb exercise ten repetition for each exercise three times per week.
  3) Flexibility Exercise : Curl up exercise and Seat and reach up exercises exercise ten repetition for each exercise three times per week.
  Lateral flexibility exercises for ten repetition for each exercise three times per week,for 12 weeks
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): Antiaging diet instructions
  Interventions: Other: aerobic exercises
- intervention group (Experimental): 1. aerobic exercises: walking :30 min on treadmill 30min at least three times per week for 12 weeks
  2. Muscle strength Exercises:
     For upper extremity : hand grip exercise, arm flexion exercise ten repetition for each exercise three times per week.
     Theraband exercises for upper limb exercise ten repetition for each exercise three times per week.
  3. Flexibility Exercise :
  Curl up exercise and Seat and reach up exercises exercise ten repetition for each exercise three times per week.
  Lateral flexibility exercises for ten repetition for each exercise three times per week,for 12 weeks and anti aging diet instruction
  Interventions: Other: aerobic exercises

INTERVENTIONS:
Other: aerobic exercises — Antiaging diet instruction :Be aware of the amount of calories, Reduce overall fat and sugar intake, Drink at least 10 glasses of water every day in order to remain healthy.
  d. Eat a variety of complex carbohydrates and vegetables instead of bread, rice, and corn.
  Other Names: flexibility exercises; strengthening exercises; anti aging diet instruction

SUMMARY:
Aging is an important fact to consider from the woman's health perspective. One of the most significant stages of aging is menopause, in which involves physical, psychological, and social changes in life

DETAILED DESCRIPTION:
This study will be carried on forty perimenopausal women. They were selected randomly from outpatient clinic of El Kaser El-Einy University Hospital, Cairo University, their age ranged from 40 to 50 years.

Group A ( Control group):

It consisted of 20 perimenopausal women. They received anti-aging diet instructions.

Group B ( Experimental group):

It will be consisted of 20 perimenopausal women.They received anti-aging therapy (Aerobic, Flexibility and strengthening exercises) with anti aging diet instructions.

Randomization:

Randomization of sample selection was achieved using closed envelop way. Classification of the sample by simple random way into two groups equal in number, twenty for each group by using forty closed envelop, each twenty envelop contained a name of a group from the two groups (Group A) or (Group B) and asking each woman to choose one envelop from them, each woman attended to the group according the name of the group written in her envelop.

ELIGIBILITY:
Inclusion Criteria:

* They complaining from fatigue, hot flushes and irregular period.
* Their Body Mass Index (BMI) between 25 to 30 .
* Their age ranged from 40 to 50 years old.
* The assessment procedures will be conducted on the same time of the day pre/post treatment.

Exclusion Criteria:

* Women with comorbidities such as cardiac disease and chest diseases as pulmonary fibrosis.
* Women received medications that might affect the neuromuscular functions at least three months before or during the study course.
* Women suffered from mental or psychological disorders.
* Women suffered from inflammatory diseases such as rheumatoid arthritis or polymyalgia rheumatic.
* Women complaining from osteoporosis.

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
6-minute walking test | 12 weeks
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
toe touch test | 12 weeks
  This test measures the flexibility of the lower back and hamstrings, and is a valid measure of this.The toe touch test is a common test of flexibility, and is an easy and quick test to perform. If using the standard testing procedure, there is a lot of published data to use for comparison.
hand held dynamometer | 12 weeks
  Hand held dynamometer demonstrated an excellent intra- and inter-rater reliability for assessment of isometric lumbar muscles strength of healthy subject at clinical setting as it is simple to use, portable and cost-effective for the precise measurement.
body composition analysis | 12 weeks
  Body composition is a method of describing what the body is made of. It includes fat, protein, minerals and body water. It also describes weight more accurately than BMI. Body composition analysis can accurately show changes in fat mass, muscle mass, and body fat percentage. This can help validate services

CONTACTS AND LOCATIONS:
Overall Officials: Amel Yousef, Study Chair — Cairo University
Locations (1):
- faculty of physical therapy, Cairo University, Giza, Egypt